CLINICAL TRIAL: NCT03620474
Title: Phase I / IIa Clinical Trial for Patients With Hepatitis C or B Virus Derived Liver Cirrhosis by CBP / β Catenin Inhibitor PRI-724
Brief Title: Safety and Effectiveness of PRI-724 for Hepatitis C or B Virus Derived Liver Cirrhosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kiminori Kimura, MD (Other)
Collaborators: Prism Pharma Co., Ltd. (Industry); Kyushu University (Other); National Center for Global Health and Medicine, Japan (Other Government); Japan Agency for Medical Research and Development (Other Government); Ohara Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Kiminori Kimura, MD, Head, Department of Hepatology, Komagome Hospital
Organization: Komagome Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRI-724-2101; UMIN000033369 (Registry Identifier: UMIN (University Hospital Medical Information) CTR)
Record Dates: First submitted 2018-07-13; First posted 2018-08-08 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Hepatitis C; Hepatitis B; Liver Cirrhoses
Keywords: Hepatitis C virus; Hepatitis B virus; liver Cirrhosis
MeSH Terms: conditions — Hepatitis C; Hepatitis B; Liver Cirrhosis | interventions — ICG 001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRI-724 (Experimental): Dose: 140, 280, 380 mg / m 2/4 hr
  Administration method:
  【Phase I Phase】 (Level 1) 140 mg / m 2/4 hr (Level 2) 280 mg / m 2/4 hr (Level 3) 380 mg / m 2/4 hr Twice weekly, continuous 4-hour intravenous administration (tolerance of administration time: ± 15 minutes). This is one cycle and 12 cycles (12 weeks in total) are carried out. However, in Phase I phase, single dose is administered on Day - 7 (tolerance: - 7 days).
  【Phase IIa phase】 Continuous intravenous administration for 4 hours twice a week at the recommended dose determined in Phase I. This is one cycle and 12 cycles (12 weeks in total) are carried out.
  Interventions: Drug: PRI-724

INTERVENTIONS:
Drug: PRI-724 — twice a week for 4 hours continuous intravenous administration of PRI-724
  Other Names: CBP-b-catenin inhibitor

SUMMARY:
To investigate the safety and efficacy of PRI-724 against HCV or HBV liver cirrhosis.

DETAILED DESCRIPTION:
【Phase I Phase】 To evaluate safety and pharmacokinetics when PRI-724 is administered to patients with HCV or HBV liver cirrhosis , and determine the recommended dose of PRI-724.

【Phase IIa phase】 To evaluate the efficacy and safety of the recommended dose of PRI-724 administered to patients with HCV or HBV liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis caused by HCV or HBV that satisfies the following (1) or (2) and satisfies (3)

  1. Patients with serum HCV-RNA positive or HCV antibody positive
  2. Patients with serum HBV-DNA positive or HBs antigen positive
  3. confirmed liver cirrhosis by liver biopsy performed in the screening period patients who received diagnosis
* Patients with Child-Pugh classification in A or B status
* Patients who satisfy HCV cirrhosis from (1) to (3), HBV cirrhosis (4) In the case of HCV cirrhosis;

  1. Patients who have not reached SVR * with DAA therapy
  2. Patients who are difficult to implement DAA therapy
  3. Patients who have been over 24 weeks after achieving SVR * with DAA therapy In case of HBV cirrhosis;
  4. Patients who have been at least 24 weeks since the start of administration of Nucleotide analogue * SVR is SVR 12 (sustained virological response at 12 weeks after the end of administration).
* Patients with Performance Status 0 to 2
* Patients aged 20 years or over and under 75 when acquiring informed consent
* Regarding participation in this trial (including liver biopsy), patients who obtained informed consent by their own voluntary intention

Exclusion Criteria:

* Patients with HCV and HBV co-infection, patients who came to cirrhosis due to causes other than HCV or HBV, or patients whose cause of cirrhosis is unknown
* Patients with esophageal gastric varices determined to be treated by endoscopic examination at screening
* Patients with complication or previous history of primary liver cancer (excluding those who have had more than one year of hepatocarcinoma resection / radiofrequency ablation)
* Merger of malignant tumor or past patients (within 3 years before screening). However, the following diseases are excluded: treated basal cell carcinoma, treated lung intraepithelial carcinoma, treated cervical carcinoma, or control superficial (not invasive) bladder carcinoma
* Patients who can not be denied HIV, HTLV-1 or syphilis
* Serum creatinine value: Patients with more than 1.5 times the upper limit of the facility reference value
* Patients with poor control of diabetes, hypertension or heart failure
* Patients with psychiatric diseases judged to have the potential to influence the implementation of clinical trials
* Patients who have severe allergy to or contrast media
* Patients with HCV who have not passed the following period after treatment for HCV cirrhosis at registration.

  * 12 weeks after the final administration of interferon
  * 16 weeks after final administration of Ribavirin
  * 16 weeks after final administration of DAA
* Patients whose dosage regimen was changed within 12 weeks prior to enrollment
* Patients who have history of drug or alcohol intoxication within 5 years before acquiring informed consent or who have history of drug or alcohol abuse within the past year
* Patients who participated in other clinical trials and clinical trials within 30 days prior to acquisition of consent, patients who used investigational drugs or investigational equipment
* Patients who received liver transplantation or other organ transplantation (including bone marrow transplantation) and patients who are difficult to intravenously administer
* Patients whose liver biopsy is expected to be difficult to perform
* Patients who are pregnant or nursing, or who are likely to become pregnant
* Male patients who do not obtain consent to contraception from the time of acquiring informed consent until the end of 12 weeks after the administration of investigational drug
* In addition, patients investigated by investigators or clinical trial doctors as judged unsuitable for this trial

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Serious side effect expression rate | 12 weeks after administration
  (Phase I)Serious side effect expression rate
liver tissue fibrosis area ratio by liver biopsy | 12 weeks after administration
  (Phase II) Amount of change from the baseline in liver tissue fibrosis area ratio by liver biopsy at 12 weeks after administration

SECONDARY OUTCOMES:
Adverse Event Expression Ratio | 12 weeks after administration
  Adverse Event Expression Ratio after PRI-724 treatment
Percentage of occurrence of side effects | 12 weeks after administration
  Percentage of occurrence of side effects after PRI-724 treatment
Pharmacokinetic parameter | 12 weeks after administration
  Maximum Plasma Concentration (Cmax)
liver stiffness from Fibro Scan | 12 weeks after administration
  Amount of change from measurement of liver stiffness by baseline from Fibro Scan at 12 weeks after administration
Child Pugh score | 12 weeks after administration
  Amount of change from baseline of Child-Pugh Score at 12 weeks after administration Child Pugh score (scale range 5-15) is obtained by adding the score for each parameter (encephalopathy, ascites, bilirubin, albumin, PT or INR).
MELD score | 12 weeks after administration
  Amount of change from baseline for MELD score at 12 weeks after administration
  The Model for End-Stage Liver Disease (MELD) is a scoring system for assessing the severity of chronic liver disease and uses the subject's values for total bilirubin, serum creatinine, and the international normalized ratio (INR) for prothrombin time to predict survival. MELD is calculated according to the following formula:
  MELD = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43
modified Histological Activity Index (HAI) by liver biopsy | 12 weeks after administration
  Change amount from baseline of modified Histological Activity Index (HAI) by liver biopsy at 12 weeks after administration

OTHER OUTCOMES:
Serum fibrosis marker level(s) | 12 weeks after administration
  Changes of level
Ascitic fluid level | 12 weeks after administration
  Changes of level

CONTACTS AND LOCATIONS:
Overall Officials: Kiminori Kimura, MD, Principal Investigator — Komagome Hospital
Locations (3):
- Japan (3):
  - Kohnodai Hospital, National Center for Global Health and Medicine, Ichikawa, Chiba
  - Tokyo Metropolitan Komagome Hospital, Bunkyō-Ku, Tokyo
  - Kyushu University Hospital, Fukuoka

REFERENCES:
- [Derived] Kimura K, Kanto T, Shimoda S, Harada K, Kimura M, Nishikawa K, Imamura J, Ogawa E, Saio M, Ikura Y, Okusaka T, Inoue K, Ishikawa T, Ieiri I, Kishimoto J, Todaka K, Kamisawa T. Safety, tolerability, and anti-fibrotic efficacy of the CBP/beta-catenin inhibitor PRI-724 in patients with hepatitis C and B virus-induced liver cirrhosis: An investigator-initiated, open-label, non-randomised, multicentre, phase 1/2a study. EBioMedicine. 2022 Jun;80:104069. doi: 10.1016/j.ebiom.2022.104069. Epub 2022 May 20. PMID 35605429